CLINICAL TRIAL: NCT00557544
Title: Randomized Controlled Trial on the Effectiveness of Metoclopramide Alone or in Combination With Ketoprofen in Acute Migraine of Child
Brief Title: Trial on Metoclopramide and Ketoprofen in Acute Migraine of Childhood
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rc 32/07
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Migraine
Keywords: migraine; metoclopramide; ketoprofen; child
MeSH Terms: conditions — Migraine Disorders | interventions — Metoclopramide; Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): metoclopramide 0,15 mg/kg and Ketoprofen 1 mg/Kg per os in single dose
  Interventions: Drug: metoclopramide; Drug: ketoprofen
- 2 (Active Comparator): metoclopramide 0,15 mg/Kg + placebo per os
  Interventions: Drug: metoclopramide; Drug: placebo
- 3 (Active Comparator): ketoprofen 1 mg/Kg and placebo in single dose
  Interventions: Drug: placebo; Drug: ketoprofen

INTERVENTIONS:
Drug: metoclopramide — metoclopramide 0,15 mg/kg
  Arms: 1; 2
Drug: placebo — placebo per os
  Arms: 2; 3
Drug: ketoprofen — ketoprofen 1 mg/Kg
  Arms: 1; 3

SUMMARY:
This is a Randomized double blind trial with the aim to estimate the effectiveness of 3 therapeutic regimes per os on migraine pain:

* metoclopramide 0,15 mg/kg + placebo
* metoclopramide 0,15 mg/Kg + ketoprofen 1 mg/kg
* ketoprofen 1 mg/Kg + placebo

Intensity of pain will be measured with linear 1-10 scale or analogic McGrath type scale every 20 min.

The main objective is the evaluation of healing times from pain in the 3 groups

ELIGIBILITY:
Inclusion Criteria:

* Children 6-17 years old with migraine presenting in emergency room

Exclusion Criteria:

* Informed consensus not obtained
* Occurring migraine still treated
* Hemiplegic migraine

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
evaluation of healing times from pain in the 3 groups | 2 hours

SECONDARY OUTCOMES:
comparison of percentage of healing from acute migraine and of relapses of pain in the three arms of trial | 2 and 24 hours respectively
need of a rescue drug for lack of effect in every arms of the trial | 2 hours and 24 hours for relapses

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Guglia, MD, Principal Investigator — IRCCS Burlo Garofolo
Locations (1):
- Edoardo Guglia, Trieste, Italy